CLINICAL TRIAL: NCT04491474
Title: Comparison of Great Occipital Nerve and Supraorbital Nerve Blockade Treatment Methods Individually and in Combination With Placebo in an Acute Migraine Attack in the Emergency Department, a Prospective, Double Blind, Randomized Controlled Study
Brief Title: Comparison of Great Occipital Nerve and Supraorbital Nerve Blockade Methods at Treatment of Acute Migraine Attack in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nihat Mujdat Hokenek, Emergency Medicine Specialist, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/514/169/20
Record Dates: First submitted 2020-07-17; First posted 2020-07-29 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Migraine Disorders
Keywords: migraine attack, nerve blockade, emergency medicine
MeSH Terms: conditions — Migraine Disorders | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Active Comparator): bilateral great occipital nerve blockade and bilateral isotonic injection into the supraorbital region.
  Interventions: Drug: Lidocaine Hydrochloride
- Group 2 (Active Comparator): bilateral supraorbital nerve blockade and bilateral isotonic injection into the great occipital nerve region
  Interventions: Drug: Lidocaine Hydrochloride
- Group 3 (Active Comparator): bilateral great occipital nerve blockade and bilateral supraorbital nerve blockade
  Interventions: Drug: Lidocaine Hydrochloride
- Group 4 (Sham Comparator): saline injection to bilateral great occipital nerve and supraorbital nerve region
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — While performing these procedures, 1 ml of 2% lidocaine hydrochloride and 1 ml of %0.9 saline will be used for creating a solution of 2 ml of 1% lidocaine for nerve block. Also 2 ml of saline will be used for placebo effect. For blocking the GON region 0.75 ml of 1% lidocaine will be applied and 0.75 ml of saline for placebo effect(8). During applying to the SON region 0.25 ml of 1% lidocaine for blockage and 0.25 ml of saline for placebo effect will be used(8). The GON injection site was planned to be 2 cm lateral and 2 cm below the occipital protrusion and the SON injection site was planned as the area with frontal incisor in the orbital arch
  Arms: Group 1; Group 2; Group 3
Drug: Placebo — There will be injection of %0.9 saline to bilaterally great occipital nerve and to bilaterally supraorbital nerve.
  Arms: Group 4

SUMMARY:
Aim Acute migraine attack is a clinical condition that is frequently encountered in emergency departments and varies from patient to patient in terms of treatment modalities. There are many different treatments whose effectiveness has been proven by concrete evidence(1). Drug treatments applied to patients are generally given intravenously or intramuscularly. Non-steroidal anti-inflammatory drugs, metoclopramide and intravenous magnesium therapy is generally used for treatment in emergency departments (1). The effectiveness of supraorbital nerve blockade and great occipital nerve blockade in migraine treatment and prophylaxis has been proven in many studies(2-6). The aim of this study is to discuss the effectiveness of supraorbital and great occipital nerve blockade treatments in acute migraine attack, when combined or used individually.

DETAILED DESCRIPTION:
Study Design The study was designed as a double-blind, prospective, randomized controlled clinical trial.

First of all patients who meet the International Headache Society (IHS CLASSIFICATION ICHD-3) migraine with or without aura criteria will be included to the study (7). Secondary it is mandatory to meet our inclusion criteria, and not to include exclusion criteria, with written informed consent to be in the study. The study will be carried out with 160 patients.

Patients who meet these conditions will be randomly divided into 4 groups. First group bilateral GON blockade and bilateral isotonic injection into the SON region,second group bilateral SON blockade and bilateral isotonic injection into the GON region,Group 3 bilateral GON blockade and bilateral SON blockade and last investigators planned to give bilateral GON and SON region saline injection to group 4.

While performing these procedures, 1 ml of 2% lidocaine and 1 ml of saline will be used for 2 ml of 1% lidocaine for nerve block. Also 2 ml of saline will be used for placebo effect. For blocking the GON region 0.75 ml of 1% lidocaine will be applied and 0.75 ml of saline for placebo effect(8). During applying to the SON region 0.25 ml of 1% lidocaine for blockage and 0.25 ml of saline for placebo effect will be used(8). The GON injection site was planned to be 2 cm lateral and 2 cm below the occipital protrusion and the SON injection site was planned as the area with frontal incisor in the orbital arch (8).

Patients will be followed up in the emergency room for 120 minutes. In the study, 1 large box will be used to ensure double blindness and randomization. There will be 2 more small boxes in it. Small boxes will be named as '' G '' and '' S '' containing the names of the nerve regions. There will be 8 injectors in each small box. There will be 8 syringes in each small box, 4 of them containing saline and 4 contains 1% lidocaine. The injectors will be numbered with the name of the box in which they are located (such as G1, G2… G8 or S1, S2… S8). In the study, 8 patients will be treated daily. In the following days, injector numbers will be written as numbers in progress (such as G9, G10..G16 and S9, S10… S16). The contents of these injectors prepared by the pharmacist will also be recorded by the pharmacist. Envelopes with random number injector combinations will be offered to patients. The combination in the envelope chosen by the patient will be applied. Injector numbers will be recorded to the data form. When the study is finished, these numbers will be checked and it will be determined which patient is given which treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting the criteria of International Headache Society (IHS CLASSIFICATION ICHD-3) migraine criteria with or without aura
2. Not taking medication before applying to the hospital
3. Over 18 years
4. Under 50 years
5. Patients with a history of migraine
6. The number of migraine attacks per month should be between 2 and 8
7. Having a headache-free period of at least 48 hours between migraine attacks
8. Diagnosis of migraine at least 1 year ago
9. Migraine prophylaxis is finished and the last dose should be taken 1 month or more

Exclusion Criteria:

1. Pregnancy
2. Epilepsy, History of Arrhythmia
3. Implantation in the skull, Cardiac pacemaker
4. Patients with a brain tumor or in an acute cerebrovascular accident clinic
5. Patients with a history of head injury
6. Past medical history of psychiatric illness
7. Patients with a fever> 38, Patients with suspected meningitis
8. Patients with acute changes of consciousness or signs of meningeal irritation
9. Hypertension (Patients with Blood Pressure> 160/110)
10. Headaches due to excessive drug use
11. Patients with headache> 15 days monthly

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Comparison of great occipital nerve and supraorbital nerve blockade methods at treatment of acute migraine attack in the emergency department, a prospective randomized controlled double blind study | 0-30th minute- 60th minute-120th minute visual analog scale pain measurements.
  VAS (Visual Analog Scale) with 100mm length, which writes start and end points, will be used as the pain assessment scale. In this scale, 0 shows the lightest pain in the form of a straight line and 100 mm indicates the most pain. This scale will be described to the participant and asked to mark the intensity of pain on the line.
  VAS values of the participants for 0 minutes, 30 minutes, 60 minutes and 120 minutes will be taken and evaluated separately. If there is no relief in the pain of the participants at the 30th minute, it is planned to administer meperidine (0.75 mcg / kg) as in similar studies as a recovery therapy(4). These patients will then be excluded from the study. Participants will be discharged after 120 minutes if they express that their pain has passed or they do not need more analgesics.

SECONDARY OUTCOMES:
Pain assessment according to Likert type verbal scale | 0 minute and 120th minute
  Secondary the participants will be asked about their responses to treatment with a scoring method from 1 to 5 according to Likert-type verbal scale, which is a verbal assessment method at 0 and 120 minutes of treatment. On this scale, they will be asked to say 1: I have a lot of pain, 2: I have a pain, 3: moderate relief, 4: I am good, 5: I am very good, and they will be asked to choose a number to evaluate their pain. This will also be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr. Lutfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
İf there is reasonable requests, I can share that time to support investigations about nerve blockade.
Supporting Information: Study Protocol, SAP
Time Frame: 5 year
Access Criteria: There should be at least 1 study about migraine attacks or nerve blockade.

REFERENCES:
- [Background] Ruiz Pinero M, Mulero Carrillo P, Pedraza Hueso MI, de la Cruz Rodriguez C, Lopez Mesonero L, Guerrero Peral AL. Pericranial nerve blockade as a preventive treatment for migraine: Experience in 60 patients. Neurologia. 2016 Sep;31(7):445-51. doi: 10.1016/j.nrl.2014.10.001. Epub 2014 Dec 24. English, Spanish. PMID 25543956
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Result] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Result] Ashkenazi A, Levin M. Greater occipital nerve block for migraine and other headaches: is it useful? Curr Pain Headache Rep. 2007 Jun;11(3):231-5. doi: 10.1007/s11916-007-0195-3. PMID 17504651
- [Result] Young W, Cook B, Malik S, Shaw J, Oshinsky M. The first 5 minutes after greater occipital nerve block. Headache. 2008 Jul;48(7):1126-8. doi: 10.1111/j.1526-4610.2008.01146.x. Epub 2008 Jun 28. PMID 18549410
- [Result] Govindappagari S, Grossman TB, Dayal AK, Grosberg BM, Vollbracht S, Robbins MS. Peripheral nerve blocks in the treatment of migraine in pregnancy. Obstet Gynecol. 2014 Dec;124(6):1169-1174. doi: 10.1097/AOG.0000000000000555. PMID 25415168
- [Result] Okmen K, Dagistan Y, Dagistan E, Kaplan N, Cancan E. Efficacy of the greater occipital nerve block in recurrent migraine type headaches. Neurol Neurochir Pol. 2016;50(3):151-4. doi: 10.1016/j.pjnns.2016.01.015. Epub 2016 Feb 6. PMID 27154440
- [Result] Ozer D, Boluk C, Turk Boru U, Altun D, Tasdemir M, Koseoglu Toksoy C. Greater occipital and supraorbital nerve blockade for the preventive treatment of migraine: a single-blind, randomized, placebo-controlled study. Curr Med Res Opin. 2019 May;35(5):909-915. doi: 10.1080/03007995.2018.1532403. Epub 2018 Oct 31. PMID 30285507
- [Result] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019 May;39(6):687-710. doi: 10.1177/0333102419828967. Epub 2019 Feb 26. PMID 30806518